CLINICAL TRIAL: NCT03820219
Title: A Pilot Study Comparing Incisional Negative Pressure Wound Therapy (Prevena) to Conventional Sterile Dressing in Patients Undergoing Thoracolumbar Posterior Spine Surgery
Brief Title: Incisional Negative Pressure Wound Therapy in Patients Undergoing Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB1023961
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2019-02

CONDITIONS: Surgical Site Infection
Keywords: spine; surgical dressing; negative pressure therapy; surgical infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: Consenting patients will be randomized to receive either standard sterile wound dressing or the Prevena™ System at the time of closure of the surgical wound.
Masking Description: The treatment allocation will be hidden for the purposes of analysis. It will be impossible to blind physicians or participants to the treatment group given the obvious difference in appearance of the Prevena™ System versus standard wound dressing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard sterile wound dressing (Placebo Comparator): Standard wound care involves the application of an occlusive dressing in the operating room, a dressing change on Post-operative Day 3 and then dressing changes as needed until suture/staple removal on Post-operative Day 14.
  Interventions: Other: Standard sterile wound dressing
- Prevena™ system (Active Comparator): The Prevena™ System is indicated for use over clean, closed incisions that continue to drain following sutured or stapled closure. It acts by removing exudate, helping hold the edges of the incision together, protecting the surgical site from external contamination in a clean, protected postoperative wound environment, until it is removed at Post-Operative Day 7.
  Interventions: Device: Prevena™ system

INTERVENTIONS:
Device: Prevena™ system — The Prevena™ System acts by removing exudate from a clean, closed incision. It helps hold the edges of the incision together, protecting the surgical site from external contamination in a clean, protected postoperative wound environment.
  Arms: Prevena™ system
Other: Standard sterile wound dressing — Standard wound care involves the application of an occlusive dressing in the operating room.
  Arms: Standard sterile wound dressing

SUMMARY:
Introduction: Posterior post-operative spine wounds involving surgery at multiple levels are known to have higher rates of wound complications relative to other areas of the body. Instrumentation, repeat surgery and prior radiation all contribute to more hostile environments for wound healing. The purpose of this study is to determine whether incisional vacuum dressings can help improve the healing/complication rates associated with these wounds.

Methods: Patients will be recruited over a two year span as part of the initial pilot study to determine the capabilities/practicality of recruitment locally. Patients will be followed in and out of hospital for 3 months or until the wound has healed clinically. The primary outcome, surgical site infection (SSI), will be evaluated using prior Centre for Disease Control (CDC) definitions. STATA will be used for statistical analysis.

Anticipated results: Although the incisional vacuum system (PrevenaTM) has been used previously for spine wounds, there are no randomized control trials compared with standard dressings. Since the infection rate in these wounds has been founds previously to be quite high (10-25%) a reduction could have profound significant benefits on patient morbidity and overall costs to the healthcare system. The pilot study will help inform the direction of a larger, potentially multi-centered trial.

Conclusion: If a large treatment effect is demonstrated with the PrevenaTM System then this could potentially change the standard of care for complex spine wounds.

DETAILED DESCRIPTION:
Patients with surgical site infection (SSI) of the spine have higher morbidity and mortality and higher costs of care. Hospital length of stay has been shown to be significantly longer, and readmission rate significantly higher, for infected patients than that for uninfected patients. Repeated surgery, typically irrigation and debridement (I&D), due to deep SSI is required in the majority of these patients. The risk of post-operative spinal wound infection is reported to be 1-20% depending on patient factors, surgical factors and spine pathology factors. The risk of SSI can be as high as 10-25% in major risk groups, such as posterior surgical approach in revision lumbar surgery, thoracolumbar trauma with neurological deficit, and in surgery for metastatic disease. Wound complications such as seroma or dehiscence can be as high as 40% in spine oncology patients, especially if they have received radiation and/or chemotherapy. Definitive management is based on etiology, clinical course, and patient risk factors. A patient who develops a post-operative wound infection often requires prolonged hospitalization, revision surgical procedures, and long-term intravenous antibiotics, which significantly increase health care resource utilization, and thus the overall cost. Awareness of risk factors and development of preventive measures can lead to improved outcomes.

There are many supplemental treatment strategies for post-operative spine infection and wound complications in addition to I&D. Vacuum assisted closure (VAC) of infected spine wounds has proven to be an acceptable adjunct to aid in the closure or staging of complex spinal wounds. The VAC system has proven to be safe and effective in the treatment of complex spinal wounds, spinal SSI and wounds that are at high risk for failed primary closure. Indications for VAC treatment as a means of preventing wound complications are evolving. Preemptive use of VAC treatment on closed primary wounds has been employed in high risk (morbidly obese) patients with acetabular fractures, and successful outcomes have been achieved. Use of VAC treatment on closed wounds as a preventive measure in properly selected patients appears safe and has effectively decreased wound complication rates. This mode of prophylactic treatment is called "incisional VAC therapy".

KCI (the manufacturer of a Vacuum Assisted Closure System) has gained FDA and Health Canada approval for a specific device called "Prevena™", which is designed for incisional vacuum therapy. The Prevena™ System is indicated for use over clean, closed incisions that continue to drain following sutured or stapled closure. It acts by removing exudate, helping hold the edges of the incision together and protecting the surgical site from external contamination in a clean, protected postoperative wound environment.

To date, no studies have been done to establish the efficacy of the Prevena™ System for use on patients requiring spine surgery to reduce wound complications such as SSI, wound dehiscence, or seroma formation. A recent systematic review of published studies examining the use of dressings and drains in posterior spinal surgery found no evidence to support the use of any particular system. A number of recent studies have also examined the incidence of surgical site infection in different high-risk populations (10-25%) and a predictive model for the development of a complex post surgical wound infection. The factors identified lead to considerable disability, cost and additional utilization of health care resources. If a prophylactic wound treatment can decrease wound complications in high risk patients, this may lead to a decreased need for post-operative services, reduced complication rate, less antibiotic usage and fewer returns to the operating room. If patients can avoid complications, they can resume normal activities faster and ultimately should have higher satisfaction.

In an era where health expenditure is literally exploding and becoming non-sustainable in many countries, cost effectiveness analysis is required to responsibly manage scarce health care resources. Specifically in the context of SSI, is the added cost of the Prevena™ System justified by the potential decrease in wound complication rate?

HYPOTHESIS:

Use of the Prevena™ System will decrease the rate of acute post-operative Surgical Site Infection.

STUDY DESIGN:

Consenting patients will be randomized to receive either standard sterile wound dressing or the Prevena™ System at the time of closure of the surgical wound. Consenting and randomization will be performed by a member of the research team. Post-stratification randomization will be performed based on the three clinical presentation groups (revision surgery, metastatic tumor and trauma with deficit). This ensures that the investigators get appropriate randomization within each of the three clinical groups.

DATA COLLECTION:

The following data elements (with their time of collection) will be collected from the patient's hospital chart of during follow-up clinical assessment

Patient Factors:

Gender (Consent) Age (Consent) Diabetes (Admission) BMI (Admission) Previous radiation to planned surgical site (Admission) Currently undergoing chemotherapy (Admission) Smoker (Admission)

Surgical Factors:

Date of Surgery (Surgery) Surgical Skin Preparation (Surgery) Estimated blood loss (Surgery) Incision size (Surgery) Drains (Surgery) Instrumentation (Surgery) Number of levels in decompression/fusion (Surgery) Blood transfusion (Surgery) Type of incision closure - staples/suture (Surgery) Procedure details - Spine Surgical Invasiveness Index (Surgery)

Hospital Stay:

Admission Date (Admission) Discharge Date (Discharge) ICU admission pre-op (Admission) ICU admission post-op (Admission) Antibiotic Use (Discharge)

Wound:

Exudate (Follow-up) Erythema (Follow-up) Separation of deep tissues (Follow-up)

Dressing Factors:

Dressing Supply Utilization (Discharge)

Data for each patient will be collected using the patient's hospital chart and visual inspection of the wound by a clinician. One questionnaire, the EQ5D, will be completed by study participants, with the help of a research assistant at Baseline (after obtaining consent), on Post-operative Day 7, Day 14 and Week 6. Participants will also be asked to complete this questionnaire if they have any unscheduled/unplanned encounters related to the occurrence of either a primary (SSI) or secondary (dehiscence/seroma) outcome during the study period.

METHODOLOGY:

Elective patients (revision and some metastatic cases) will be introduced to the study at the time of surgical consent by a member of the research team. Emergent patients (all trauma and most metastatic cases) will be introduced to the study pre-operatively in the Emergency Department or in the Orthopaedic Clinic by a member of the research team. Study participants will be randomized prior to surgery to receive either the Prevena™ System or standard wound care.

All consenting participants will be randomized, based on the three primary diagnostic groups (revision surgery, metastatic disease or fracture with deficit). Study participants who receive the 'standard wound care' will have the dressing changed 3 days after their surgery and will have study encounters on Post-operative Day 7, Day 14 and Week 6 for wound inspection, dressing change (Day 7) and suture/staple removal (Day 14). Study participants who receive the Prevena™ System will have the same schedule of study encounters for wound inspection (Post-operative Day 7, Day 14 and Week 6). The Prevena™ System will be removed on Day 7 and a dry, sterile dressing will be applied. On Day 14 sutures/staples will be removed.

Patients who have not yet been discharged at the time of the scheduled study encounter will be seen in hospital. Patients who have been discharged prior to any scheduled study encounters will be seen in a follow-up spine clinic.

Participants will all be assigned a unique study ID and the treatment allocation will be hidden for the purposes of analysis. It will be impossible to blind physicians or participants to the treatment group given the obvious difference in appearance of the Prevena™ System versus standard wound dressing.

STATISTICS:

A power calculation has been performed to determine the number of participants required. This analysis has presumed an incidence of SSI of 15% (based on an averaging calculation of published data for these high risk groups), and used a 2-tailed analysis, assuming a power of 0.8 and a Type I error of 5%. For a 50% decrease in primary outcome rates, Surgical Site Infection, (15% to 7.5%), 275 participants per group will be required. The pilot data generated from the proposed study will allow for refinement of this target recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Capable of and agree to consent to randomization
* Require spine surgery with a posterior midline incision that involves the thoracic, lumbar and/or sacral spine
* Be one of the following clinical presentation groups:

  1. Metastatic Tumor of the Thoracic or Lumbar spine (T1-S5), requiring instrumentation and decompression, with or without pre-operative site radiation
  2. Revisions Surgery requiring additional instrumentation or revision instrumentation, for thoracolumbar degeneration or deformity (T1-S1), index surgery >6 months prior
  3. Acute Traumatic Thoracolumbar (T1-L5) fracture(s) with neurological deficit (AIS A-C), requiring instrumentation and decompression

Exclusion Criteria:

Initially:

* Undergoing percutaneous surgery
* Active Surgical Site infection or Primary Spinal Column infection or Distant Site Infection (urinary tract, respiratory tract, etc.)

Subsequently:

* Failure to complete the 6-week clinical follow-up (Loss to Follow Up)
* Second surgery, at the same anatomical site, required during study time period (six weeks), for causes other than primary (SSI) or secondary (Dehiscence, Seroma) study endpoints.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Rate of acute post-operative Surgical Site Infection (SSI) | 6 weeks
  The incidence rate of SSI for patients with the Prevena™ System will be compared to those with the standard dressing.

SECONDARY OUTCOMES:
Post operative wound seroma or dehiscence | 1 week
  The incidence of wounds requiring aspiration, surgical exploration, or incision repair for patients with the Prevena™ System will be compared to those with the standard dressing.
Resource time commitment | 2 weeks
  The time and resource commitment for post-operative, in-hospital, wound management for patients with the Prevena™ System will be compared to those with the standard dressing. This data is collected on a standardized log sheet appended to the nursing folio.
Return visits | 6 weeks
  The number of unanticipated post-op clinic visits, hospital readmissions and, emergency department/urgent-unplanned clinic evaluations for patients with the Prevena™ System will be compared to those with the standard dressing.

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Health, Halifax, Nova Scotia (NS), Canada